CLINICAL TRIAL: NCT06087380
Title: The Effectiveness of Auricular Acupressure on Improving Pain and Heart Variability in Patients After Cervical Spine Surgery
Brief Title: Auricular Acupressure on Improving Pain and Heart Variability in Patients After Cervical Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Liu-ying Yin, National Taipei University of Nursing and Health Sciences, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021-09-008B
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Auricular Acupressure; Cervical Spine Surgery
Keywords: cervical spine surgery; post-operative pain; auricular acupressure; heart variability.
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arms and Interventions (Experimental): The experimental group A total of 32 patients to undergo auricular acupuncture interventional
  Interventions: Procedure: auricular acupressure; Other: standard ward care
- No Intervention: Control group: (Other): The control group total 30 patients No interventions implemented
  Interventions: Other: standard ward care

INTERVENTIONS:
Procedure: auricular acupressure — Auricular pressure The experimental group commenced auricular acupressure intervention post-surgery. Questionnaire assessments and heart rate variability measurements were conducted in the experimental group on the first, second, third, and fourth days before discharge.
  Arms: Arms and Interventions
Other: standard ward care — standard ward care

SUMMARY:
The primary objective of this study is to investigate the effectiveness of auricular acupressure in improving post-cervical spine surgery pain and heart rate variability in patients.

DETAILED DESCRIPTION:
This study adopts a quasi-experimental research design, where a medical center in northern Taiwan served as the enrollment location. Both the experimental group and the control group received standard ward care. The experimental group commenced auricular acupressure intervention post-surgery. Questionnaire assessments and heart rate variability measurements were conducted in the experimental group on the first, second, third, and fourth days before discharge. The control group did not receive auricular acupressure and underwent only questionnaire assessments and heart rate variability testing. Measurement tools included the McGill Pain Questionnaire and the Heart Master wrist-worn physiological monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Those who are over 20 years old and have undergone cervical spine surgery.
2. Those who have clear consciousness and can communicate in Mandarin or Taiwanese.
3. Patients who have undergone cervical spine surgery and have no complications (such as wound infection or postoperative limb mobility impairment) disability).
4. Those who are willing to cooperate with ear acupuncture and heart rate variability testing.
5. Those who agree to participate in the research and sign the consent form.
6. The skin of the auricle is intact and has no deformation, defects or allergies.-

Exclusion Criteria:

1. Those who use self-controlled pain control (PCA) after surgery.
2. Those diagnosed with mental illness or cognitive impairment.
3. Those who are transferred to the intensive care unit after surgery.
4. Those who use breathing aids.
5. Those with major chronic diseases, such as cardiovascular disease or cancer.
6. Those who develop delirium after surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
short-form Questionnaire McGill Pain, SF-MPQ) | post op 1-4 day
  It mainly assesses the nature and intensity of pain. The scale is mainly divided into three parts. The first part is the pain level index, which includes 11 questions on the sensory level of pain experience and 4 questions on the emotional level of pain experience, a total of 15 questions. The higher the score, the greater the pain. The more serious it is; the second part is the current pain intensity, the higher the score, the more severe the pain; the third part is the visual analog scale (VAS), the higher the score, the more severe the pain.

SECONDARY OUTCOMES:
Heart Rhythm Master Wrist Physiological Monitor | post op 1-4 day
  Monitors spectrum values such as high frequency of heart rate variability, low frequency of heart rate variability, and power ratio of high and low frequency of heart rate variability.The standard values of its measurement parameters: high-frequency power parameter (HF) is 40-60%, low-frequency power parameter (LF) is 40-60%, and autonomic nervous system activity balance parameter (LF/HF) is 0.8-1.5 ms2.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yin Liu, Master, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Taipei veterans general hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No